CLINICAL TRIAL: NCT06476301
Title: Efficacy and Safety of Rivaroxaban in the Early Postoperative Period for Patients With Bioprosthetic Valves: A Prospective, Randomized, Controlled Non-Inferiority Trial
Brief Title: Efficacy and Safety of Rivaroxaban in the Early Postoperative Period for Patients With Bioprosthetic Valves
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT-2023-0325
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Anticoagulation
Keywords: warfarin; rivaroxaban; Bioprosthetic valve; anticoagulation
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warfarin group (No Intervention): A 3-6-month anticoagulation therapy with warfarin is recommended after the BPV surgery. Patients allocated to the warfarin group will adhere to a target INR range of 2 to 3. Patients 65 > years old and low weight should take warfarin 2.5mg/day and all other patients should take 5mg/day. During hospitalization, the INR will be reassessed daily, and regular measurements (at least every four weeks) should be conducted post-discharge to ensure ongoing patient stability.
- rivaroxaban group (Experimental): Patients allocated to the rivaroxaban group will be administered a dose of 20 mg orally once daily (to be taken with food), or 15 mg once daily in patients with moderate renal impairment at screening (defined as creatinine clearance rate, CrCl between 30 and 49 mL/min).
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — To compare the efficacy and safety of rivaroxaban as an early anticoagulant therapy for BPV patients with the traditional postoperative anticoagulant warfarin
  Arms: rivaroxaban group

SUMMARY:
this study aims to comprehensively evaluate the efficacy and safety profiles of rivaroxaban and warfarin during the initial postoperative period following surgical bioprosthetic valve in patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* Patients who underwent successful surgical bioprosthetic valve replacement or repair to either the mitral, aortic position or both
* Signed informed consent

Exclusion Criteria:

* Aged below 18 or over 80 years
* Mechanical heart valves (MHV)
* Bioprosthetic valve transcatheter valve replacement (TAVR)
* Hemorrhage risk-related criteria

  1. Active internal bleeding
  2. Major surgical procedure or trauma within 30 days before the randomization visit
  3. History of intracranial, intraocular, spinal, gastrointestinal, or atraumatic intra-articular bleeding
  4. Chronic hemorrhagic disorder
  5. Planned invasive procedure with potential for uncontrolled bleeding, including major surgery
* Concomitant conditions and therapies

  1. Clinically overt stroke within the past 3 months
  2. Major surgery within 1 month
  3. Acute coronary syndrome within 1 month
  4. Active infective endocarditis
  5. Severe hepatic impairment、hepatic disease associated with coagulopathy or Moderate and severe hepatic impairment (Child-Pugh Class B or C)
  6. Uncontrolled severe hypertension
  7. Active malignancy
* Medication-related

  1. Hypersensitivity or contraindications to Rivaroxaban, VKA, heparin.
  2. Concomitant treatment with strong inhibitors of both CYP3A4 and P-gp (e.g., azole antifungals, such as ketoconazole and itraconazole, or HIV protease inhibitors, such as ritonavir)
  3. Concomitant treatment with strong inducers of CYP3A4 (e.g., carbamazepine, phenytoin, rifampin, etc.)
* HAS-BLED score>3
* Others

  1. Abnormal local laboratory results, such as Platelet count < 50 x109/L、Hemoglobin < 8 g/dL (5 mmol/L)
  2. Female subjects of childbearing potential without using adequate contraception、
  3. Female pregnant or breast-feeding
  4. Participation is not likely to comply with the study procedures or will complete follow-up
  5. Participation in another clinical trial that potentially interferes with the current study
  6. Life expectancy less than 6 months beyond the targeted last visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 0.5, 1, 3, and 6 months
  Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.
Major cardiovascular events (stroke, transient ischemic attack (TIA), valve thrombosis, systemic embolism not related to the central nervous system (CNS), hospitalization due to heart failure) | 0.5, 1, 3, and 6 months
  Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.
Major bleeding | 0.5, 1, 3, and 6 months
  Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.

SECONDARY OUTCOMES:
Thromboembolic events (stroke, TIA, deep venous thrombosis, pulmonary embolism, non-CNS systemic embolism, valve thrombosis). | 0.5, 1, 3, and 6 months
  The Efficacy endpoint was defined as the composite of death from cardiovascular causes or Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.
Cardiovascular causes death | 0.5, 1, 3, and 6 months
  Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.
Major bleeding events and clinically relevant non-major (CRNM) bleeding events and minor bleeding events | 0.5, 1, 3, and 6 months
  Patients will be scheduled for outpatient clinic or phone visits at intervals of 0.5, 1, 3, and 6 months following enrollment. During these visits, patients will be instructed to document any symptoms indicative of clinical thromboembolic or bleeding events. If such symptoms are reported, patients may undergo necessary diagnostic and laboratory testing. Cardiac CT and transthoracic echocardiography will be conducted at the 3-month and 6-month marks post-randomization.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Zhang C, Pan MM, Lin HW, Xue S, Xie B, Gu ZC. Design and rationale of the multicenter randomized clinical trial (REVERSE): Efficacy and safety of rivaroxaban in the early postoperative period for patients with bioprosthetic valve replacement or valve repair. Int J Cardiol. 2025 Apr 15;425:133023. doi: 10.1016/j.ijcard.2025.133023. Epub 2025 Feb 1. PMID 39900192